CLINICAL TRIAL: NCT04932044
Title: Construction and Longitudinal Following Up the Effects of Early Sleep Facilitation Program on Preterm Infants' Sleep, Health After Discharge, and Caregiver's Sleep, Stress, Quality of Life, and Attachment
Brief Title: Sleep Program on Preterm Infants' Sleep, and Caregiver's Sleep, Stress, Quality of Life, and Attachment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Defense Medical Center, Taiwan (Other)
Responsible Party: Principal Investigator, Hsiang-Yun Lan, Assistant Professor, National Defense Medical Center, Taiwan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: C202005014
Record Dates: First submitted 2021-05-28; First posted 2021-06-18 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-06

CONDITIONS: Preterm Infants; Sleep; Quality of Life
Keywords: Preterm Infants; Sleep; Quality of Life; Attachment; Actigraphy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early Sleep Facilitation Program (Experimental): Perform sleep circadian rhythm training during hospitalization, and provide caregivers with nursing guidance to promote sleep of premature infants before discharge
  Interventions: Behavioral: Early Sleep Facilitation Program; Other: Routine care
- routine care and provide general discharge care and nursing guidance (Active Comparator): Routine care and provide general discharge care and nursing guidance.
  Interventions: Other: Routine care

INTERVENTIONS:
Behavioral: Early Sleep Facilitation Program — It is divided into two stages. The first stage is to provide sleep circadian rhythm training for preterm infants during hospitalization, and the second stage is to give the caregiver the nursing guidance to promote preterm infants' sleep before preterm infants discharged from the hospital. Moreover, continue to give nursing guidance and follow its implementation status within two months after discharge.
  Arms: Early Sleep Facilitation Program
Other: Routine care — Receives routine care and provide general discharge care and nursing guidance.

SUMMARY:
This research plan to construct an "Early Sleep Facilitation Program"and to explore the effects of the "early sleep Facilitation program" on the sleep and health of preterm infants and the sleep, stress, quality of life and attachment of the caregiver for a Long-term follow-up research.

The proposed study has six specific aims:

1. Explore the effect of "Early Sleep Facilitation Program" on the sleep of preterm infants during hospitalization and after returning home.
2. Explore the effect of "Early Sleep Facilitation Program" on the health of preterm infants during hospitalization and after returning home.
3. Explore the effect of "Early Sleep Facilitation Program" on the sleep of the caregiver after preterm infants during hospitalization and after returning home.
4. Explore the effect of the "Early Sleep Facilitation Program" on the stress of the caregivers of preterm infants during hospitalization and after returning home.
5. Explore the effect of "Early Sleep Facilitation Program" on the quality of life of the caregivers of preterm infants during hospitalization and after returning home.
6. Explore the effect of "Early Sleep Facilitation Program" on the attachment of the caregivers of preterm infants during hospitalization and after returning home.

DETAILED DESCRIPTION:
Background and purpose:

Preterm infants need to receive intensive care in a neonatal intensive care unit (NICU) to survive, but the sleep of preterm infants is disturbed by the environment of the intensive care unit, invasive treatment and care activities. When a preterm infant's sleep is interrupted, it not only affects his physical growth, behavior and emotional development, but also affects his recovery from illness and the length of hospital stay, and even affects his sleep quality and development after returning home. However, medical personnel are busy with clinical practice, seldom pay attention to the sleep development of preterm infants. In the past, few studies paid attention to the factors that affect the sleep of preterm infants after returning home, and few studies also explored the sleep and physical and mental health of preterm infants and their main caregivers after returning home. Sleep intervention in preterm infants was mostly a single outcome indicator; besides, past studies lacked objective sleep instruments and long-term follow-up studies.

Based on the above research gaps, this research plan to construct an "early sleep Facilitation program" and to explore the effects of the "Early Sleep Facilitation Program" on the sleep and health of preterm infants and the sleep, stress, quality of life and attachment of the caregiver for a Long-term follow-up research.

The proposed study has six specific aims:

1. Explore the effect of "Early Sleep Facilitation Program" on the sleep of preterm infants during hospitalization and after returning home.
2. Explore the effect of "Early Sleep Facilitation Program" on the health of preterm infants during hospitalization and after returning home.
3. Explore the effect of "Early Sleep Facilitation Program" on the sleep of the caregiver after preterm infants during hospitalization and after returning home.
4. Explore the effect of the "Early Sleep Facilitation Program" on the stress of the caregivers of preterm infants during hospitalization and after returning home.
5. Explore the effect of "Early Sleep Facilitation Program" on the quality of life of the caregivers of preterm infants during hospitalization and after returning home.
6. Explore the effect of "Early Sleep Facilitation Program" on the attachment of the caregivers of preterm infants during hospitalization and after returning home.

Methods:

This randomized controlled trial will adopt a longitudinal repeated measures design to examine the " Early Sleep Facilitation Program " on the sleep and health of preterm infants and the sleep, stress, quality of life and attachment of the caregiver. Preterm infants and the caregiver were recruited by convenience sampling in Neonatal Intensive Care Unit and Infant Intermediate Care Unit of a medical center in northern Taiwan from July in 2020 to December in 2022. There are two different intervention modes (intervention group and control group), the intervention group receives " Early Sleep Facilitation Program " and the control group receives routine care. The program is divided into two stages. The first stage is to provide sleep circadian rhythm training for preterm infants during hospitalization, and the second stage is to give the caregiver the nursing guidance to promote preterm infants' sleep before preterm infants discharged from the hospital. Moreover, continue to give nursing guidance and follow its implementation status after the first month and the second month after discharge. The control group receives routine care and provide general discharge care and nursing guidance. The questionnaires and physiological measurements will be used to collect the data. The two groups will collect data during hospitalization, one week before discharge, and the first month and the second month after discharge. We will use generalized estimation equations method to analyze research data.

ELIGIBILITY:
Inclusion Criteria:

1. Preterm infants gestational age (GA) > 28 weeks and < 37 weeks, and birth weight less than 2200 grams;
2. The main caregiver of the preterm infants can communicate in Mandarin and Taiwanese;
3. The parents of the preterm infants and their main caregivers agrees to participate in this research and signs the research consent form

Exclusion Criteria:

1. Premature infant is diagnosed with limb dysfunction or brain neuropathy, such as: third or fourth degree intraventricular hemorrhage or peripheral ventricular leukomalacia;
2. Other diseases that affect sleep, such as: congenital nerve development Abnormalities, epilepsy;
3. Those who need to take muscle relaxants, sedatives or bronchodilators

Ages: 28 Weeks to 37 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 70 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Preterm Infants' Sleep- Actigraphy -T1 | T1-baseline collect preterm infants after 32 weeks of gestation before intervention
  Accessed by Actigraphy
Preterm Infants' Sleep- Actigraphy -T2 | T2- preterm infants one week before discharge
  Accessed by Actigraphy
Preterm Infants' Sleep- Actigraphy -T3 | T3- preterm infants the first month after discharge
  Accessed by Actigraphy
Preterm Infants' Sleep- Actigraphy -T4 | T4- preterm infants second month after discharge
  Accessed by Actigraphy
Preterm Infants' Sleep- sleep log -T1 | T1-baseline collect preterm infants after 32 weeks of gestation before intervention
  The primary caregiver records the sleep log of premature babies. The sleep log is used to understand the total sleep hours of premature infants, the number of awake hours/times at night, sleep efficiency, and factors that may interfere with sleep.
Preterm Infants' Sleep- sleep log -T2 | T2- preterm infants one week before discharge
  The primary caregiver records the sleep log of premature babies. The sleep log is used to understand the total sleep hours of premature infants, the number of awake hours/times at night, sleep efficiency, and factors that may interfere with sleep.
Preterm Infants' Sleep- sleep log -T3 | T3- preterm infants the first month after discharge
  The primary caregiver records the sleep log of premature babies. The sleep log is used to understand the total sleep hours of premature infants, the number of awake hours/times at night, sleep efficiency, and factors that may interfere with sleep.
Preterm Infants' Sleep- sleep log -T4 | T4- preterm infants second month after discharge
  The primary caregiver records the sleep log of premature babies. The sleep log is used to understand the total sleep hours of premature infants, the number of awake hours/times at night, sleep efficiency, and factors that may interfere with sleep.
Preterm Infants' Health- Health Assessment Form-weight-T1 | T1-baseline collect preterm infants after 32 weeks of gestation before intervention
  The weight is measured by the researcher with a baby weight scale. This device record data: weight(kg).
  Health Assessment Form for premature infants information included anthropometric measurements: size at weight (kg), head circumference (cm), and recumbent length (cm) with the new World Health Organization (WHO) Growth Standard for a growth chart. Calculate Growth curve and Growth percentage.
Preterm Infants' Health- Health Assessment Form-weight-T2 | T2- preterm infants one week before discharge
  The weight is measured by the researcher with a baby weight scale. This device record data: weight(kg).
  Health Assessment Form for premature infants information included anthropometric measurements: size at weight (kg), head circumference (cm), and recumbent length (cm) with the new World Health Organization (WHO) Growth Standard for a growth chart. Calculate Growth curve and Growth percentage.
Preterm Infants' Health- Health Assessment Form-weight-T3 | T3- preterm infants the first month after discharge
  The weight is measured by the researcher with a baby weight scale. This device record data: weight(kg).
  Health Assessment Form for premature infants information included anthropometric measurements: size at weight (kg), head circumference (cm), and recumbent length (cm) with the new World Health Organization (WHO) Growth Standard for a growth chart. Calculate Growth curve and Growth percentage.
Preterm Infants' Health- Health Assessment Form-weight-T4 | T4- preterm infants second month after discharge
  The weight is measured by the researcher with a baby weight scale. This device record data: weight(kg).
  Health Assessment Form for premature infants information included anthropometric measurements: size at weight (kg), head circumference (cm), and recumbent length (cm) with the new World Health Organization (WHO) Growth Standard for a growth chart. Calculate Growth curve and Growth percentage.
Preterm Infants' Health- Health Assessment Form- head circumference-T1 | T1-baseline collect preterm infants after 32 weeks of gestation before intervention
  The head circumference is measured by the researcher with tape measure. This device record data: head circumference (cm).
  Health Assessment Form for premature infants information included anthropometric measurements: size at weight (kg), head circumference (cm), and recumbent length (cm) with the new World Health Organization (WHO) Growth Standard for a growth chart. Calculate Growth curve and Growth percentage.
Preterm Infants' Health- Health Assessment Form- head circumference-T2 | T2- preterm infants one week before discharge
  The head circumference is measured by the researcher with tape measure. This device record data: head circumference (cm).
  Health Assessment Form for premature infants information included anthropometric measurements: size at weight (kg), head circumference (cm), and recumbent length (cm) with the new World Health Organization (WHO) Growth Standard for a growth chart. Calculate Growth curve and Growth percentage.
Preterm Infants' Health- Health Assessment Form- head circumference-T3 | T3- preterm infants the first month after discharge
  The head circumference is measured by the researcher with tape measure. This device record data: head circumference (cm).
  Health Assessment Form for premature infants information included anthropometric measurements: size at weight (kg), head circumference (cm), and recumbent length (cm) with the new World Health Organization (WHO) Growth Standard for a growth chart. Calculate Growth curve and Growth percentage.
Preterm Infants' Health- Health Assessment Form- head circumference-T4 | T4- preterm infants second month after discharge
  The head circumference is measured by the researcher with tape measure. This device record data: head circumference (cm).
  Health Assessment Form for premature infants information included anthropometric measurements: size at weight (kg), head circumference (cm), and recumbent length (cm) with the new World Health Organization (WHO) Growth Standard for a growth chart. Calculate Growth curve and Growth percentage.
Preterm Infants' Health- Nutrition data-T1 | T1-baseline collect preterm infants after 32 weeks of gestation before intervention
  Data on nutrition support included: recordings of types of feeding (breast milk or formula), total fluid intakes, and number of feeding interruptions.
Preterm Infants' Health- Nutrition data-T2 | T2- preterm infants one week before discharge
  Data on nutrition support included: recordings of types of feeding (breast milk or formula), total fluid intakes, and number of feeding interruptions.
Preterm Infants' Health- Nutrition data-T3 | T3- preterm infants the first month after discharge
  Data on nutrition support included: recordings of types of feeding (breast milk or formula), total fluid intakes, and number of feeding interruptions.
Preterm Infants' Health- Nutrition data-T4 | T4- preterm infants second month after discharge
  Data on nutrition support included: recordings of types of feeding (breast milk or formula), total fluid intakes, and number of feeding interruptions.
Caregivers' Sleep- Actigraphy-T1 | T1-baseline collect Caregiver of preterm infants after 32 weeks of gestation before intervention
  Accessed by Actigraphy. Actigraphy is a validated method of objectively measuring sleep parameters and average motor activity.
Caregivers' Sleep- Actigraphy-T2 | T2- preterm infants one week before discharge
  Accessed by Actigraphy. Actigraphy is a validated method of objectively measuring sleep parameters and average motor activity.
Caregivers' Sleep- Actigraphy-T3 | T3- preterm infants the first month after discharge
  Accessed by Actigraphy. Actigraphy is a validated method of objectively measuring sleep parameters and average motor activity.
Caregivers' Sleep- Actigraphy-T4 | T4- preterm infants second month after discharge
  Accessed by Actigraphy. Actigraphy is a validated method of objectively measuring sleep parameters and average motor activity.
Caregivers' Sleep- Pittsburgh Sleep Quality Index (PSQI)-T1 | T1-baseline collect Caregiver of preterm infants after 32 weeks of gestation before intervention
  The Pittsburgh Sleep Quality Index (PSQI) is a self-report questionnaire that assesses sleep quality over a 1-month time interval. The measure consists of 19 items, the PSQI measures several different aspects of sleep, offering seven component scores and one composite score. The component scores consist of subjective sleep quality, sleep latency (i.e., how long it takes to fall asleep), sleep duration, habitual sleep efficiency (i.e., the percentage of time in bed that one is asleep), sleep disturbances, use of sleeping medication, and daytime dysfunction.
Caregivers' Sleep- Pittsburgh Sleep Quality Index (PSQI)-T2 | T2- preterm infants one week before discharge
  The Pittsburgh Sleep Quality Index (PSQI) is a self-report questionnaire that assesses sleep quality over a 1-month time interval. The measure consists of 19 items, the PSQI measures several different aspects of sleep, offering seven component scores and one composite score. The component scores consist of subjective sleep quality, sleep latency (i.e., how long it takes to fall asleep), sleep duration, habitual sleep efficiency (i.e., the percentage of time in bed that one is asleep), sleep disturbances, use of sleeping medication, and daytime dysfunction.
Caregivers' Sleep- Pittsburgh Sleep Quality Index (PSQI)-T3 | T3- preterm infants the first month after discharge
  The Pittsburgh Sleep Quality Index (PSQI) is a self-report questionnaire that assesses sleep quality over a 1-month time interval. The measure consists of 19 items, the PSQI measures several different aspects of sleep, offering seven component scores and one composite score. The component scores consist of subjective sleep quality, sleep latency (i.e., how long it takes to fall asleep), sleep duration, habitual sleep efficiency (i.e., the percentage of time in bed that one is asleep), sleep disturbances, use of sleeping medication, and daytime dysfunction.
Caregivers' Sleep- Pittsburgh Sleep Quality Index (PSQI)-T4 | T4- preterm infants second month after discharge
  The Pittsburgh Sleep Quality Index (PSQI) is a self-report questionnaire that assesses sleep quality over a 1-month time interval. The measure consists of 19 items, the PSQI measures several different aspects of sleep, offering seven component scores and one composite score. The component scores consist of subjective sleep quality, sleep latency (i.e., how long it takes to fall asleep), sleep duration, habitual sleep efficiency (i.e., the percentage of time in bed that one is asleep), sleep disturbances, use of sleeping medication, and daytime dysfunction.
Caregivers' Sleep- Sleep log-T1 | T1-baseline collect Caregiver of preterm infants after 32 weeks of gestation before intervention
  Sleep log: record the sleep time and sleep status of the previous day to understand the total sleep hours, the number of awake hours/times at night, sleep efficiency, and whether there are events that affect the mood of falling asleep, medication or physical discomfort, whether to consume irritating substances and alcohol, etc. And use a scale of 1 to 5 points to assess the quality of sleep the night before and the level of wakefulness when waking up.
Caregivers' Sleep- Sleep log-T2 | T2- preterm infants one week before discharge
  Sleep log: record the sleep time and sleep status of the previous day to understand the total sleep hours, the number of awake hours/times at night, sleep efficiency, and whether there are events that affect the mood of falling asleep, medication or physical discomfort, whether to consume irritating substances and alcohol, etc. And use a scale of 1 to 5 points to assess the quality of sleep the night before and the level of wakefulness when waking up.
Caregivers' Sleep- Sleep log-T3 | T3- preterm infants the first month after discharge
  Sleep log: record the sleep time and sleep status of the previous day to understand the total sleep hours, the number of awake hours/times at night, sleep efficiency, and whether there are events that affect the mood of falling asleep, medication or physical discomfort, whether to consume irritating substances and alcohol, etc. And use a scale of 1 to 5 points to assess the quality of sleep the night before and the level of wakefulness when waking up.
Caregivers' Sleep- Sleep log-T4 | T4- preterm infants second month after discharge
  Sleep log: record the sleep time and sleep status of the previous day to understand the total sleep hours, the number of awake hours/times at night, sleep efficiency, and whether there are events that affect the mood of falling asleep, medication or physical discomfort, whether to consume irritating substances and alcohol, etc. And use a scale of 1 to 5 points to assess the quality of sleep the night before and the level of wakefulness when waking up.
Caregivers' Stress- T1 | T1-baseline collect Caregiver of preterm infants after 32 weeks of gestation before intervention
  Parenting Stress Index-Third Edition short form (PSI-SF) The PSI Short Form is a direct derivative of the full-length test and consists of a 36-item self-scoring questionnaire/profile. Each question is based on Likert's five-point. The total score is between 36-180 points, the higher the score, the greater the parental pressure.
Caregivers' Stress- T2 | T2- preterm infants one week before discharge
  Parenting Stress Index-Third Edition short form (PSI-SF) The PSI Short Form is a direct derivative of the full-length test and consists of a 36-item self-scoring questionnaire/profile. Each question is based on Likert's five-point. The total score is between 36-180 points, the higher the score, the greater the parental pressure.
Caregivers' Stress- T3 | T3- preterm infants the first month after discharge
  Parenting Stress Index-Third Edition short form (PSI-SF) The PSI Short Form is a direct derivative of the full-length test and consists of a 36-item self-scoring questionnaire/profile. Each question is based on Likert's five-point. The total score is between 36-180 points, the higher the score, the greater the parental pressure.
Caregivers' Stress- T4 | T4- preterm infants second month after discharge
  Parenting Stress Index-Third Edition short form (PSI-SF) The PSI Short Form is a direct derivative of the full-length test and consists of a 36-item self-scoring questionnaire/profile. Each question is based on Likert's five-point. The total score is between 36-180 points, the higher the score, the greater the parental pressure.
Caregivers' quality of life-T1 | T1-baseline collect Caregiver of preterm infants after 32 weeks of gestation before intervention
  World Health Organization Quality of Life-BREF (WHOQOL-BREF) The WHOQOL is a quality of life assessment developed by the WHOQOL Group with fifteen international field centres, simultaneously, in an attempt to develop a quality of life assessment that would be applicable cross-culturally. There are 28 questions in the questionnaire. The content includes four aspects: physical health, psychology, social relations and environment. Each question is based on Likert's five-point. The higher the score, the better the quality of life.
Caregivers' quality of life-T2 | T2- preterm infants one week before discharge
  World Health Organization Quality of Life-BREF (WHOQOL-BREF) The WHOQOL is a quality of life assessment developed by the WHOQOL Group with fifteen international field centres, simultaneously, in an attempt to develop a quality of life assessment that would be applicable cross-culturally. There are 28 questions in the questionnaire. The content includes four aspects: physical health, psychology, social relations and environment. Each question is based on Likert's five-point. The higher the score, the better the quality of life.
Caregivers' quality of life-T3 | T3- preterm infants the first month after discharge
  World Health Organization Quality of Life-BREF (WHOQOL-BREF) The WHOQOL is a quality of life assessment developed by the WHOQOL Group with fifteen international field centres, simultaneously, in an attempt to develop a quality of life assessment that would be applicable cross-culturally. There are 28 questions in the questionnaire. The content includes four aspects: physical health, psychology, social relations and environment. Each question is based on Likert's five-point. The higher the score, the better the quality of life.
Caregivers' quality of life-T4 | T4- preterm infants second month after discharge
  World Health Organization Quality of Life-BREF (WHOQOL-BREF) The WHOQOL is a quality of life assessment developed by the WHOQOL Group with fifteen international field centres, simultaneously, in an attempt to develop a quality of life assessment that would be applicable cross-culturally. There are 28 questions in the questionnaire. The content includes four aspects: physical health, psychology, social relations and environment. Each question is based on Likert's five-point. The higher the score, the better the quality of life.
Caregivers' attachment-T1 | T1-baseline collect Caregiver of preterm infants after 32 weeks of gestation before intervention
  Maternal Attachment Inventory (MAI) The Maternal Attachment Inventory(MAI) has 26 questions on the scale. The questions use a response level of 1 to 4. The 1 point means almost none, 2 points means occasionally, 3 points means often, and 4 points means almost often.
  The higher the total score, the closer the maternal-infant attachment.
Caregivers' attachment-T2 | T2- preterm infants one week before discharge
  Maternal Attachment Inventory (MAI) The Maternal Attachment Inventory(MAI) has 26 questions on the scale. The questions use a response level of 1 to 4. The 1 point means almost none, 2 points means occasionally, 3 points means often, and 4 points means almost often.
  The higher the total score, the closer the maternal-infant attachment.
Caregivers' attachment-T3 | T3- preterm infants the first month after discharge
  Maternal Attachment Inventory (MAI) The Maternal Attachment Inventory(MAI) has 26 questions on the scale. The questions use a response level of 1 to 4. The 1 point means almost none, 2 points means occasionally, 3 points means often, and 4 points means almost often.
  The higher the total score, the closer the maternal-infant attachment.
Caregivers' attachment-T4 | T4- preterm infants second month after discharge
  Maternal Attachment Inventory (MAI) The Maternal Attachment Inventory(MAI) has 26 questions on the scale. The questions use a response level of 1 to 4. The 1 point means almost none, 2 points means occasionally, 3 points means often, and 4 points means almost often.
  The higher the total score, the closer the maternal-infant attachment.

CONTACTS AND LOCATIONS:
Overall Officials: Hsiang-Yun Lan, Asst. Prof., Principal Investigator — National Defense Medical Center, Taiwan
Locations (1):
- National defense medical center, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No